CLINICAL TRIAL: NCT07338695
Title: Evaluation of Hemodynamic Changes in Peripheral Microcirculation in Response to Photobiomodulation Using Non-Invasive Optical and Thermal Technologies
Brief Title: The Effect of Photobiomodulation on Microvascular Blood Flow: The Role of Wavelength and Skin Temperature
Acronym: PBM&MBF01
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Afeka, The Tel-Aviv Academic College of Engineering (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 09-12-2024-AFK; PBM&MBF01 (Other: Afeka)
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Microcirculation
Keywords: Photoniomodulation; low-level laser; microcirculatory blood flow

STUDY DESIGN:
Intervention Model Description: This is a within-subject crossover study in which participants receive photobiomodulation at blue and near-infrared wavelengths in separate sessions, with the order of exposure assigned in a crossover manner. Participants may present with functional peripheral vasoconstriction or normal peripheral temperature at baseline; these baseline characteristics will be used for subgroup analyses and do not define separate study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Blue → Near-Infrared PBM (Experimental): Participants receive photobiomodulation at a blue wavelength in the first session and at a near-infrared wavelength in the second session.
  Interventions: Device: Photobiomodulation - Blue Wavelength; Device: Photobiomodulation - Near Infrared
- Near-Infrared → Blue PBM (Experimental): Participants receive photobiomodulation at a near-infrared wavelength in the first session and at a blue wavelength in the second session.
  Interventions: Device: Photobiomodulation - Blue Wavelength; Device: Photobiomodulation - Near Infrared

INTERVENTIONS:
Device: Photobiomodulation - Blue Wavelength — Photobiomodulation delivered at a blue wavelength (400-500 nm) to the hands during a single study session as part of a randomized crossover design.
Device: Photobiomodulation - Near Infrared — Photobiomodulation delivered at a near-infrared wavelength (780-1100 nm) to the hands during a single study session as part of a randomized crossover design.

SUMMARY:
The objective of this study is to assess peripheral microcirculatory hemodynamic responses to photobiomodulation in participants with normal circulation and with functional peripheral vasoconstriction, using noninvasive thermography, photoplethysmography, and laser Doppler flowmetry.

DETAILED DESCRIPTION:
This is a within-subject experimental study in which each participant completes two study sessions. Microvascular and systemic variables are continuously monitored in response to photobiomodulation delivered at either a blue or near-infrared wavelength, with each wavelength applied in a separate session.

Each session includes a baseline period with controlled breathing, followed by photobiomodulation and a 20-minute post-intervention follow-up period. Peripheral microcirculatory responses are assessed using noninvasive thermography, photoplethysmography, and laser Doppler flowmetry.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, between 20 and 75 years of age.
2. Willing to sign informed consent.
3. Willing to participate in two separate sessions, one for each wavelength.
4. Able to avoid caffeine and alcohol for at least 3 hours before each session.
5. Able to sit comfortably with both hands at heart level for the full measurement duration.

Exclusion Criteria:

1. Currently smoking
2. Any abnormal skin condition in the area of light irradiation.
3. Pregnant, having given birth less than 3 months ago, and/or breastfeeding.
4. History of photosensitive conditions or use of photosensitizing medications
5. Suffering from significant concurrent illness, such as cardiac disorders or pertinent neurological disorders.
6. As per the Investigator's discretion, any physical or mental condition that might make it unsafe for the subject to participate in this study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Capillary blood flow | Up to 1 hour
  Capillary blood flow, expressed as red blood cell flux (perfusion units), measured continuously using laser Doppler flowmetry (≥10 Hz sampling rate) from baseline through the end of each study session.

SECONDARY OUTCOMES:
Temperature distribution over hands measured by thermography | Up to 1 hour
  Thermal images will be acquired using a FLIR infrared camera, and spatial temperature distribution over the hands will be analyzed. Images will be acquired at one-minute intervals from baseline through the end of each study session.

OTHER OUTCOMES:
Photoplethysmography (PPG)-derived perfusion response | Up to 1 hour
  Continuous photoplethysmography (PPG) will be recorded from the hand, and PPG-derived perfusion metrics (e.g., pulse amplitude and related indices) will be quantified to assess changes in peripheral microcirculation following photobiomodulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Afeka, Tel-Aviv Academic College of Engineering, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gavish L, Hoffer O, Rabin N, Halak M, Shkilevich S, Shayovitz Y, Weizman G, Haim O, Gavish B, Gertz SD, Ovadia-Blechman Z. Microcirculatory Response to Photobiomodulation-Why Some Respond and Others Do Not: A Randomized Controlled Study. Lasers Surg Med. 2020 Nov;52(9):863-872. doi: 10.1002/lsm.23225. Epub 2020 Feb 17. PMID 32064652
- [Background] Ovadia-Blechman Z, Hauptman Y, Rabin N, Wiezman G, Hoffer O, Gertz SD, Gavish B, Gavish L. Morphological features of the photoplethysmographic signal: a new approach to characterize the microcirculatory response to photobiomodulation. Front Physiol. 2023 Sep 25;14:1175470. doi: 10.3389/fphys.2023.1175470. eCollection 2023. PMID 37817983